CLINICAL TRIAL: NCT00712491
Title: A Phase 1/2, Randomized Clinical Study to Assess the Safety and Efficacy of Sirolimus in Patients With Newly Diagnosed, Treatment-Naive Sub-Foveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: Phase 1/2 Study of an Ocular Sirolimus (Rapamycin) Formulation in Patients With Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Collaborators: MacuSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMD-002
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2010-07

CONDITIONS: Age-related Macular Degeneration; Choroidal Neovascularization
Keywords: wet AMD; CNV
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sirolimus
- 2 (Experimental)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Three subconjunctival injections of 1320 micrograms sirolimus each.
  Other Names: MS-R002, rapamycin
  Arms: 1
Drug: Sirolimus — Three intravitreal injections of 352 micrograms sirolimus each.
  Other Names: MS-R001, rapamycin
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an ocular sirolimus (rapamycin) formulation via different injection routes in patients with treatment-naive sub-foveal choroidal neovascularization secondary to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria include, but are not limited to:

* Diagnosed with sub-foveal choroidal neovascularization secondary to age-related macular degeneration
* Visual acuity of 20/50 to 20/200 in study eye

Exclusion Criteria:

* Any other ocular disease that could compromise vision in the study eye
* History of any prior treatment for choroidal neovascularization in the study eye
* Presence of other causes of choroidal neovascularization other than secondary to age-related macular degeneration

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity by ETDRS | 180 days

SECONDARY OUTCOMES:
Best-corrected visual acuity by ETDRS | 60 days, 120 days
Safety across injection routes | Through 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joel Naor, MD, Study Director — MacuSight, Inc.
Locations (1):
- Retinal Consultants of Arizona, Phoenix, Arizona, United States